CLINICAL TRIAL: NCT00887549
Title: An Exploratory, Prospective Phase II Study to Investigate Progression-Free Survival, Response and Overall Survival Seen With Pemetrexed/Cisplatin and the Role of Thymidylate Synthase Expression
Brief Title: A Study of Thymidylate Synthase Expression in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13069; H3E-BP-JMIK (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2011-08-30 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed (Experimental)
  Interventions: Drug: pemetrexed; Drug: cisplatin

INTERVENTIONS:
Drug: pemetrexed — Induction Therapy: 500 milligrams per square meter (mg/m^2), intravenous, day 1 of each 21 day cycle for the first 4 cycles; Maintenance Therapy: 500 milligrams per square meter (mg/m^2), intravenous, day 1 of each 21 day cycle until progression or unacceptable toxicity occurs
  Other Names: Alimta; LY231514
Drug: cisplatin — Induction Therapy: 75 mg/m^2, intravenous, day 1 of each 21 day cycle for the first 4 cycles

SUMMARY:
Thymidylate synthase (TS) is a substance the body produces naturally. The purpose of this research is to determine if there is a link between TS production and how well patients respond to treatment of non-squamous non-small cell lung cancer (NSCLC). The aim for the future is that doctors could have a better understanding in advance about which patients might respond well to pemetrexed based on how much TS they produce.

DETAILED DESCRIPTION:
All patients on this study will receive 4 intravenous injections of the chemotherapy drugs pemetrexed and cisplatin (with each injection approximately 3 weeks apart). Patients who complete 4 such injections and respond well to their treatment may continue to receive an injection of chemotherapy drug pemetrexed (approximately every 3 weeks). In general terms, treatment will last until either the patient or the doctor decides that there is no clear benefit in continuing with the treatment.

TS levels will be measured from the tumour sample used to make the original diagnosis of NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Stage 3B or 4 Non-Small Cell Lung Cancer of the non- squamous type
* Patients must at least be able to be physically mobile, take care of yourself and be able to perform light activities such as light housework or office work
* Patients must not have had previous chemotherapy treatment for lung cancer
* Patients must not have had radiotherapy in the last 30 days
* Patients must have measureable tumor lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines or disease that can be evaluated on computed tomography (CT) scan
* Patients' test results assessing the function of their blood forming tissue, kidneys, liver and lungs are satisfactory
* Women must be sterile, postmenopausal or on contraception and men must be sterile or on contraception

Exclusion Criteria:

* Patients cannot have received other investigational drugs within the last 30 days
* Patients cannot have any serious, uncontrolled medical condition that might compromise their ability to take part in the study safely
* Patients cannot have a current second primary malignant tumor
* Patients cannot be having current treatment with any other anti-tumor therapy
* Patients cannot have had a yellow fever vaccination within 30 days of enrolment
* Patients who are unable to take vitamins (including injections of vitamin B12) or oral cortisone medication
* Patients who are unable to stop taking more than 1.3 grams of aspirin on a daily basis or non-steroidal anti-inflammatory agents
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dublin, Ireland
- United Kingdom (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Derby, Derbyshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Exeter, Devon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maidstone, Kent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Preston, Lancashire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liverpool, Merseyside
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northwood, Middlesex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scunthorpe, North Lincolnshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belfast, Northern Ireland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nottingham, Nottinghamshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aberdeen, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wolverhampton, West Midlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grimsby
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester

REFERENCES:
- [Derived] Fennell DA, Myrand SP, Nguyen TS, Ferry D, Kerr KM, Maxwell P, Moore SD, Visseren-Grul C, Das M, Nicolson MC. Association between gene expression profiles and clinical outcome of pemetrexed-based treatment in patients with advanced non-squamous non-small cell lung cancer: exploratory results from a phase II study. PLoS One. 2014 Sep 24;9(9):e107455. doi: 10.1371/journal.pone.0107455. eCollection 2014. PMID 25250715

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial consists of induction therapy (up to 4 cycles of pemetrexed-cisplatin treatment) and maintenance therapy (pemetrexed only). Only participants who do not develop disease progression during induction therapy are eligible to receive maintenance therapy.
Groups:
- Pemetrexed: Induction Therapy: pemetrexed 500 milligrams per square meter (mg/m^2) and cisplatin 75 mg/m^2, intravenous, day 1 of each 21 day cycle for the first 4 cycles; Maintenance Therapy: pemetrexed 500 milligrams per square meter (mg/m^2), intravenous, day 1 of each 21 day cycle until progression or unacceptable toxicity occurs
Period: Induction Therapy
Arm/Group | Pemetrexed
Started | 70
Completed | 43
Not Completed | 27
Not completed — Adverse Event | 8
Not completed — Physician Decision | 1
Not completed — Progressive Disease | 13
Not completed — Death due to Study Disease | 4
Not completed — Death due to Study Drug Toxicity | 1
Period: Maintenance Therapy
Arm/Group | Pemetrexed
Started | 43
Completed | 0
Not Completed | 43
Not completed — Adverse Event | 16
Not completed — Physician Decision | 1
Not completed — Progressive Disease | 25
Not completed — Death due to adverse event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 70
Age Continuous [Mean (Standard Deviation); unit: years] | 63.0 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 38
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 69
  Asian | 1
Region of Enrollment [Number; unit: participants]
  Ireland | 4
  United Kingdom | 66
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0- Fully active | 24
    1- Ambulatory, Restricted Strenuous Activity | 46
Pathological Diagnosis [Number; unit: participants]
  Adenocarcinoma, not otherwise specified (NOS) | 34
  Adenocarcinoma, acinar | 1
  Adenocarcinoma, poorly differentiated | 20
  Bronchioalveolar Carcinoma | 6
  Carcinoma, Non-Small Cell, Lung (NSCL), (NOS) | 3
  Carcinoma, NSC, Poorly Differentiated, Lung | 5
  Carcinoma, undifferentiated | 1
Past and Current Tobacco Usage [Number; unit: participants]
  Never used tobacco products | 6
  Ever used tobacco products | 64

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is time from first dose to first observation of disease progression/death (any cause). PFS is reported for participants with thymidylate synthase (TS) scores. For participants not known to have died by the data cut-off date and who do not have progressive disease, PFS will be censored at date of last objective progression-free disease assessment. For participants who receive systemic anticancer therapy after study drug discontinuation and prior to disease progression/death, PFS will be censored at date of last objective progression-free disease assessment prior to chemotherapy.
Time Frame: Baseline to measured progressive disease with follow-up every 6 weeks until progression of disease (up to 18 months after the last participant commenced induction therapy)
Population: Population for the efficacy assessment includes all treated participants with a valid TS expression assessment. Six participants were censored for PFS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 60
months | 5.5 [3.9 to 6.9]
Statistical Analysis 1: Comparison: Pemetrexed; Test type: Superiority or Other; p < 0.0001, Regression, Cox; The Cox model, based upon participant level data, included PFS as dependent variable and TS score in the nucleus as independent variable; Hazard Ratio (HR) = 1.015, 95% CI 2-sided [1.008 to 1.021]

2. Secondary Outcome: Percentage of Participants With Tumor Response (Tumor Response Rate)
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors (RECIST 1.0) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria. Percentage of participants with tumor response was determined by the number of participants with PR or CR (confirmed or not) divided by the total number of treated participants multiplied by 100.
Time Frame: Baseline to disease progression (up to 20 months)
Population: All enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 70
percentage of participants | 30 [19.62 to 42.13]

3. Secondary Outcome: Percentage of Participants With Concordance Between Local and Central Histological Diagnosis
Description: A centralized pathology review on all enrolled participants was performed to confirm the histological diagnosis performed at the site. Upon review of the local diagnosis obtained at the respective site, the central reviewer established whether or not there was an agreement between the local and central diagnosis. The percentage of participants with concordance was defined as the number of participants for which there was an agreement divided by the number of treated participants (concordance rate) multiplied by 100.
Time Frame: Baseline
Population: All enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 70
percentage of participants | 78.6 [67.1 to 87.5]

4. Secondary Outcome: Percentage of Participants Surviving at 18 Months (Overall Survival Rate)
Description: The percentage of participants surviving at 18 months was defined as the number of treated participants who had not died prior to 18 months from the date of their first dose divided by the total number of treated participants multiplied by 100. For participants who are alive, overall survival was censored at the last contact.
Time Frame: Baseline to date of death (up to 24.5 months)
Population: All enrolled participants. Nineteen participants were censored for overall survival.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 70
percentage of participants | 37.1 [25.89 to 49.52]

ADVERSE EVENTS:
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 41/70
Other Adverse Events (participants affected / at risk) | 67/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=70)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 7 (7)
Chest discomfort (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Non-cardiac chest pain (General disorders) | 5 (5)
Oedema peripheral (General disorders) | 2 (3)
Pyrexia (General disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 6 (6)
Lung infection (Infections and infestations) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 2 (2)
Penile infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Vena cava injury (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 3 (3)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=70)
Anaemia (Blood and lymphatic system disorders) | 15 (15)
Neutropenia (Blood and lymphatic system disorders) | 7 (10)
Tinnitus (Ear and labyrinth disorders) | 5 (5)
Lacrimation increased (Eye disorders) | 15 (15)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 23 (28)
Diarrhoea (Gastrointestinal disorders) | 19 (23)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 10 (12)
Nausea (Gastrointestinal disorders) | 33 (53)
Stomatitis (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 25 (34)
Chest pain (General disorders) | 4 (4)
Fatigue (General disorders) | 39 (43)
Mucosal inflammation (General disorders) | 5 (5)
Oedema peripheral (General disorders) | 10 (11)
Cellulitis (Infections and infestations) | 5 (6)
Lower respiratory tract infection (Infections and infestations) | 13 (16)
Oral candidiasis (Infections and infestations) | 6 (7)
Urinary tract infection (Infections and infestations) | 4 (5)
Alanine aminotransferase increased (Investigations) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 6 (6)
Blood creatinine increased (Investigations) | 11 (11)
Creatinine renal clearance decreased (Investigations) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 4 (4)
Haemoglobin decreased (Investigations) | 10 (13)
Neutrophil count decreased (Investigations) | 6 (9)
Weight decreased (Investigations) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 22 (23)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 12 (12)
Headache (Nervous system disorders) | 13 (14)
Lethargy (Nervous system disorders) | 9 (9)
Neuropathy peripheral (Nervous system disorders) | 6 (7)
Tremor (Nervous system disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11)
Rash (Skin and subcutaneous tissue disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days